## **STATISTICAL ANALYSIS PLAN**

NCT Number: NCT01297309

Study Title: A Long-term Open-label Study Investigating the Safety and Tolerability

of NPSP558, a Recombinant Human Parathyroid Hormone (rhPTH[1-84]), for the Treatment of Adults with Hypoparathyroidism – A Clinical

Extension Study (RACE)

Study Number: PAR-C10-008

SAP Version: SAP Amendment 1

SAP Version Date: 22 March 2018

## STATISTICAL ANALYSIS PLAN

A Long Term Open-label Study Investigating the Safety and Tolerability of NPSP558, a <u>Recombinant Human Parathyroid</u> Hormone (rhPTH [1-84]), for the Treatment of Adults with Hypoparathyroidism – <u>A Clinical Extension Study (RACE)</u>

Study No. PAR-C10-008

## **Authorization Signature Page**

A Long-term Open-label Study Investigating the Safety and Tolerability of NPSP558, a Recombinant Human Parathyroid Hormone (rhPTH [1-84]), for the Treatment of Adults with Hypoparathyroidism  $-\underline{A}$  Clinical Extension Study (RACE)







## **Table of contents**

| Auth | orizatio | on Signature Page | 2 |
|---|---|---|---|
| List o | f Figur | res and Tables | 5 |
| Modi | fication | ı History | 6 |
| | | eviations and definition of terms | |
| 1. | | uction | |
| 2. | • | Objectives | |
| | 2.1. | Primary objective | |
| | 2.2. | Secondary objective | 10 |
| 3. | Study | Design | 11 |
| | 3.1. | General Description | 11 |
| | 3.2. | Treatments | |
| | | 3.2.1. Treatments Administered | |
| | 2.2 | 3.2.2. Method of Assigning Subjects | |
| | 3.3. | Determination of Sample Size | |
| | 3.4. | Changes in the Conduct of the Study or Planned Analyses | |
| | | 3.4.1. Changes in the Conduct of the Study | |
| | Ti cc | | |
| 4. | | cy and Safety Variables | |
| | 4.1. | Schedule of Evaluations and Procedures | |
| | 4.2. | Efficacy Endpoint | |
| | 4.3. | Other Efficacy Endpoints | 22 |
| | 4.4. | Exploratory Endpoints | 22 |
| | 4.5. | Safety Endpoints | 22 |
| 5. | Statist | ical Methods | 24 |
| | 5.1. | General Methodology | 24 |
| | 5.2. | Adjustments for Covariates | 24 |
| | 5.3. | Visit Windows | 24 |
| | | 5.3.1. Analysis Visit Windows | 24 |
| | | 5.3.2. Definition of Baseline | |
| | 5.4. | Handling of Dropouts or Missing Data | |
| | | 5.4.1. Handling of Dropouts or Missing Data for Efficacy Analysis | |
| | | 5.4.2. Handling of Dropouts or Missing Data for Safety Analysis | |
| | 5.5. | Interim Analyses and Data Monitoring. | |
| | 5.6. | Multicenter Studies. | |
| | 5.7. | Multiple Comparisons/Multiplicity | |
| | 5.8. | Active-Control Studies Intended to Show Non-inferiority or Equivalence | |
| | 5.9. | Examination of Subgroups | |
| 6. | Statist | ical Analysis | 28 |

| 10. | | ndix I: Summary of Changes Made to SAP version 1.0 Dated Octob | |
|---|---|---|---|
| 9. | Refer | rences | 38 |
| 8. | Mock | Tables, Listings and Graphs (TLG) | 37 |
| 7. | Progr | ramming Conventions for Outputs | 36 |
| | | 6.8.5. Concomitant Medications | 34 |
| | | 6.8.4.5. PTH and ECP Antibodies | 34 |
| | | 6.8.4.4. Physical Examination Findings | |
| | | 6.8.4.3. Serum 25-Hydroxyvitamin D and Serum 1,25-dihydroxyvitamin D | |
| | | 6.8.4.1. Vital Signs | |
| | | 6.8.4. Vital Signs, Physical Findings, and Other Observations Related to Safety. | |
| | | 6.8.3. ECG Evaluations. | 33 |
| | | 6.8.2. Clinical Laboratory Evaluation | |
| | 0.0. | 6.8.1. Adverse Events | |
| | 6.8. | Analysis of Safety | |
| | | 6.7.4. Exploratory Analyses | |
| | | 6.7.3. Subset Analyses | |
| | | 6.7.2. Other Analyses | |
| | | 6.7.1. Primary Analysis | 29 |
| | 6.7. | Analysis of Efficacy | 29 |
| | | 6.6.1. Exposure during this (RACE) study | |
| | 6.6. | Extent of Exposure | 29 |
| | 6.5. | Measurements of Treatment Compliance | 28 |
| | 6.4. | Demographic and Other Baseline Characteristics | 28 |
| | 6.3. | Analysis Populations | |
| | 6.2. | Protocol Deviations | |
| | 6.1. | 1 | 28 |

## List of Figures and Tables

| Figure 1. 1 | Study Design – First 12 Months of Study | 12 |
|---|---|---|
| Figure 1. 2 | Study Design – Long-term Extension | 12 |
| Table 4. 1 | Schedule of Evaluations and Procedures – First 12 Months of Study | 15 |
| Table 4. 2 | Schedule of Evaluations and Procedures – Long-term Extension to Month | |
| | 36 | 17 |
| Table 4. 3 | Schedule of Evaluations and Procedures – Long-term Extension after | |
| | Month 36 | 19 |
| Table 4. 4 | Schedule of Follow-up Visits and Procedures for Subjects with | |
| | PTH-specific Antibodies at Final Visit | 21 |
| Table 5. 1 | Analysis Visit Window Definition (1st 12 Month of Study) | 24 |
| Table 6. 1 | Definition of the Stages of Clcr3 | 32 |
| Table 6. 2 | Markedly Abnormal Laboratory Criteria <sup>4</sup> | 32 |
| Table 6. 3 | Potentially Clinically Significant Post-Baseline ECG <sup>5,6</sup> | 33 |
| Table 6. 4 | Markedly Abnormal Post-Baseline Vital Signs <sup>7</sup> | 34 |

## **Modification History**

| Unique<br>Identifier<br>for this<br>Version | Date of the<br>Document<br>Version | Author | Significant Changes from<br>Previous Authorized Version |
|---|---|---|---|
| Amendment 1 v2.0 | 22MAR2018 | PPD | Study design description and schedule tables were updated to be aligned with Protocol Amendment 6. |

Document: Shire PAR Author: 

## List of abbreviations and definition of terms

AE Adverse Event

AESI Adverse Event of Special Interest ALT Alanine Aminotransferase AST Aspartate Aminotransferase

ATC Anatomic Therapeutic Chemical classification

BMD Bone mineral density
BMI Body Mass Index

BSAP Bone-specific alkaline phosphatase

BUN Blood Urea Nitrogen
CBC Complete blood count
CPK Creatine phosphokinase

CTx C-terminal telopeptide of type 1 collagen
DSMB Data and Safety Monitoring Board
DXA Dual-energy x-ray absorptiometry

ECG Electrocardiogram
ECP Escherichia coli protein
EOT End of Treatment

eCRF Electronic case report form

CLcr Cockcroft-Gault Creatinine Clearance
FDA Food and Drug Administration
FSH Follicle-stimulating hormone
GFR Glomerular filtration rate

GI Gastrointestinal HR Heart Rate

ICF Informed consent form

ICH International Conference on Harmonization

ITT Intent-to-Treat

IVRInteractive Voice ResponseIWRInteractive Web ResponseLDHLactate dehydrogenase

MedDRA Medical Dictionary for Regulatory Activities

ms milliseconds

NDA New Drug Application

P1NP Procollagen amino-terminal peptide

PR In electrocardiography, the time from the beginning of the P wave (onset of

atrial depolarization) to the beginning of the QRS complex

PT Preferred Term
PTH Parathyroid hormone

QD Daily

QRS In electrocardiography, the QRS complex represents the time it takes for

depolarization of the ventricles

QT In electrocardiography, the time from the beginning of the QRS complex to

the end of the T wave

QTc QT interval corrected for heart rate

QTcB QT corrected for heart rate by the Bazett method QTcF QT corrected for heart rate by the Fridericia method

RBC Red Blood Cell

RELAY A Randomized, Dose-blinded Study to Investigate the Safety and Efficacy

of NPSP558, a Recombinant Human Parathyroid Hormone (rhPTH[1-84]),, at Fixed Doses of 25 ug and 50 ug for the Treatment of Adults With

at Fixed Doses of 25  $\mu g$  and 50  $\mu g$  for the Treatment of Adults With

Hypoparathyroidism. Study No. is PAR-C10-007

REPLACE A Randomized, Double-blind, Placebo-Controlled, Phase 3 Study to

Investigate the Use of NPSP558, a Recombinant Human Parathyroid

Hormone (rhPTH[1-84]) for the Treatment of Adults with

Hypoparathyroidism. Study No. is CL1-11-040 Recombinant human parathyroid hormone

RR In electrocardiography, the time duration between two consecutive R waves

Document: Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link

Author: 

Version Number: 2.0

Version Date: March 22, 2018

| SAE | Serious Adverse Event |
|-----|---------------------------|
| SAP | Statistical Analysis Plan |

SC Subcutaneous

SI International System of Units

SOC System Organ Class

TEAE Treatment Emergent Adverse Event
TESAE Treatment Emergent Serious Adverse Event

ULN Upper Limit of Normal WBC White Blood Cell

WHO World Health Organization

Document: Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link
Author: Version Number:

Author: Version Number: 2.0 Version Date: March 22, 2018

## 1. Introduction

This document describes the rules and conventions for data handling and methodologies for statistical analysis to be used in the presentation and analysis of efficacy and safety data for protocol PAR-C10-008 (RACE). It describes, in detail, the data and variables to be summarized and analyzed, including specifics of the statistical analyses to be performed. This statistical analysis plan is based on Protocol Amendment 6, dated October 24, 2016.

Hypoparathyroidism is a condition in which there is deficient production of parathyroid hormone (PTH) from the parathyroid glands. The deficiency of PTH results in decreased calcium reabsorption from renal tubules, malabsorption of calcium from the gastrointestinal (GI) tract and reduced calcium mobilization from bone. Hypoparathyroidism is the most common cause of chronic hypocalcemia.

NPSP558 (rhPTH[1-84]) is recombinant human parathyroid hormone that is identical in structure to endogenous human parathyroid hormone (hPTH), a single-chain polypeptide consisting of 84 amino acid residues (rhPTH[1-84]). This is a 12-month open-label study investigating the safety and tolerability of NPSP558 for the Treatment of Adults with Hypoparathyroidism.

A Phase 3 study is currently ongoing (CL1-11-040, REPLACE) to investigate the effects of daily subcutaneous (SC) injections of rhPTH[1-84] at doses of 50, 75, or 100  $\mu$ g. An 8-week study of fixed doses of 25 and 50  $\mu$ g (PAR-C10-007, RELAY) is currently being undertaken to explore a broader range of treatment dose options.

Document: Author:  Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link
PPD
Version Number:


2.0

## 2. Study Objectives

## 2.1. Primary objective

To demonstrate the long-term safety and tolerability of SC rhPTH[1-84] as hormone replacement therapy for the treatment of adult subjects with hypoparathyroidism.

## 2.2. Secondary objective

- To evaluate the impact of different preparations of calcium on the response to rhPTH[1-84] replacement therapy
- To demonstrate that dosing with rhPTH[1-84] across a dose range of 25 to 100 μg SC can be implemented in a safe and effective manner and can be maintained throughout long-term treatment
- To evaluate the impact of calcium-sparing diuretics on serum and urinary calcium

Document:
Author:


Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link
Version Number:
2.0

#### 3. **Study Design**

#### 3.1. **General Description**

This study is a long-term, open-label study using rhPTH[1-84] for the treatment of adults with hypoparathyroidism. Subjects can enroll if they either previously completed the NPSP558 RELAY study (PAR-C10-007) (8 weeks of active therapy) and/or completed the REPLACE study (CL1-11-040) (Visit 18).

The goal of this study is to optimize rhPTH[1-84] dosing while reducing calcitriol and oral calcium (carbonate or citrate) supplementation to as low as safely possible and maintaining total serum calcium levels. Dose adjustments to rhPTH[1-84] and to the calcium/calcitriol supplements and safety monitoring of calcium levels are explained in protocol Appendix 2, rhPTH[1-84] and Supplement Titration Guideline.

- The starting dose of rhPTH[1-84] for this study will be 25 or 50 µg SC once daily (OD)
- Subjects may have their rhPTH[1-84] dose adjusted by the investigator at any time during the study, with the goal of achieving or maintaining total serum calcium levels in the range of 8.0 to 9.0 mg/dL.
- If ANY predose (trough) total serum calcium is >11.9 mg/dL study drug will be stopped.
- Subjects will have blood draws to assess total serum calcium levels (which may be performed locally) 3 to 5 days after ANY dose adjustment of rhPTH[1-84], after any significant change in doses of calcium and/or calcitriol supplements, or at any other time at the discretion of the investigator.
- Study visits during the first 12 months of the study will be conducted at Weeks 1 (baseline), 4, 8, and then every 8 weeks thereafter up to Week 48 (Visit 8). The Week 52 visit (Visit 9) is scheduled 4 weeks later.
- At any time following the Week 16 (Visit 4), subjects who are on a stable dose of rhPTH[1-84] and have a 24-hour urine calcium >300 mg (males) and >250 mg (females) may be treated for hypercalciuria with calcium-sparing diuretics, if this therapy had not been introduced prior to the study.
- At the end of Week 52, subjects will be invited to extend their study drug regimen until January 2018 or after the completiong of the last patient's Month 72 visit, whichever comes laslt..
- During this time, subjects will return to the clinic for interim visits every 2 months (Months 14, 16, 18, etc).
- After the End of Treatment visit or early termination visit, subjects who will not continue rhPTH[1-84] treatment will have their total serum calcium and phosphate levels measured 3 to 5 days after the last dose of study medication. Doses of calcium and active vitamin D supplements will be adjusted by the Investigator as appropriate. Thereafter, the Investigator will repeat serum calcium/phosphate monitoring and supplement dose adjustments as appropriate to achieve target serum calcium/phosphate concentrations until the follow up phone call 4 weeks  $\pm$  7days after end of treatment visit. After the 4 weeks follow up phone call, further management of hypoparathyroidism will occur as part of the subject's long-term non-study medical care.

Document: Author:

PPD

A schematic presentation of the study design is displayed in Figure 1.1 and Figure 1.2.

Figure 1. 1 Study Design – First 12 Months of Study



Figure 1. 2 Study Design – Long-term Extension



## 3.2. Treatments

## 3.2.1. Treatments Administered

At the beginning of the study, subjects will receive rhPTH[1-84] 25 or 50  $\mu$ g SC QD in an open-label fashion. Subjects may have their rhPTH[1-84] dose adjusted upwards in increments of 25  $\mu$ g to a maximum of 100  $\mu$ g SC QD, with the goal of achieving or maintaining total serum calcium levels in the range of 8.0 to 9.0 mg/dL. The rhPTH[1-84] dose may be adjusted downward at any time as needed to maintain appropriate total serum calcium levels

Document: Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link
Author: 

Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link

(approximately 8.0 to 9.0 mg/dL) or due to any safety concerns. rhPTH[1-84] is to be administered into alternating thighs each morning via a multi-dose injection pen device.

## 3.2.2. Method of Assigning Subjects

Subjects previously enrolled in or who completed the REPLACE or RELAY studies will utilize the same 8-digit subject number that they had been assigned during that study. This number will be utilized to identify the subject throughout the study period. New subjects who were never entered into the REPLACE study will be assigned a new 8-digit subject number.

Subjects will receive study treatment in an open-label fashion at starting doses of rhPTH[1-84] 25 or 50  $\mu g$  SC QD:

- Subjects with a total serum calcium value of ≤ 9.5 mg/dL will have a starting dose of 50 μg.
- Subjects with a total serum calcium value of > 9.5 mg/dL will have a starting dose as follows:
  - Subjects who are taking supplements (≥ 500 mg oral calcium and/or any calcitriol) will have the supplements reduced or stopped and will start at a dose of 50 μg SC QD.
  - $\circ$  Subjects who are taking minimal or no supplemental calcium (< 500 mg oral calcium) and no calcitriol will have a starting dose of 25  $\mu$ g SC QD.

The kit number from which cartridges are dispensed to a subject will be recorded on the appropriate eCRF. All subsequent kit numbers will be similarly recorded. All doses of study medication for each subject must be taken from the kit(s) designated for that subject and cartridges from an assigned kit will not be dispensed to any other subject.

## 3.3. Determination of Sample Size

Approximately 50 subjects are anticipated to be enrolled. This sample size is based on an estimate of the number of subjects who potentially could roll over from RELAY and/or REPLACE study and is not calculated based on the statistical assumptions.

## 3.4. Changes in the Conduct of the Study or Planned Analyses

## 3.4.1. Changes in the Conduct of the Study

The SAP is based on Protocol Amendment 6, dated October 24, 2016. Any change of the conduct of the study will be documented in the clinical study report. Any significant changes in the planned analysis will prompt another version of the SAP and therefore a revised SAP.

## 3.4.2. Changes from Analyses Planned in the Protocol

No changes from protocol specified analyses are planned.

Document: Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link
Author: 

Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link

## 4. Efficacy and Safety Variables

## 4.1. Schedule of Evaluations and Procedures

All clinical study evaluations will be performed according to Table 6.1, Table 6.2, and Table 6.3. Details of the exact date and time of medical assessments (day/month/year) will be documented in the eCRF. Any deviations from protocol requirements will be documented in the eCRF. A schedule of follow-up visits and procedures for subjects who test positive for PTH-specific antibodies at the last visit is provided in Table 6.4.

Document: Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link
Author: PPD Version Number: 2.0

Table 4. 1 Schedule of Evaluations and Procedures – First 12 Months of Study

| Visit Number | | Int. | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Procedures / Proposed Study Week <sup>a</sup> | $\mathbf{BL^b}$ | 1 <sup>c</sup> | 4 | 8 | 16 | 24 | 32 | 40 | 48 | 52 |
| Visit Windows | ± 3 days | ± 2 days | ± 7 days | ± 7<br>days | ±7 days | ± 7 days | ± 7 days | ± 7 days | ±7 days | ± 7<br>days |
| Informed Consent | X | | | | | | | | | |
| Review Inclusion/Exclusion Criteria | X | | | | | | | | | |
| Medical History (updated from RELAY/REPLACE) | X | | | | | | | | | |
| Concomitant medications (ongoing) | X | | X | X | X | X | X | X | X | X |
| Concomitant medications (new) | X | | X | X | X | X | X | X | X | X |
| Adverse event monitoring (ongoing) | X | | X | X | X | X | X | X | X | X |
| Adverse event monitoring (new) | X | | X | X | X | X | X | X | X | X |
| Assessment of clinical episodes of hypocalcemia and hypercalcemia | X | | X | X | X | X | X | X | X | X |
| Physical examination | X | | | | | | | | | X |
| Vital signs <sup>d</sup> and weight | X | | X | X | X | X | X | X | X | X |
| Electrocardiogram (12-lead) (centrally read) | X | | | | | | | | | X |
| Bone mineral density by DXA <sup>e</sup> | X | | | | | | | | | X |
| Hematology <sup>f</sup> | X | | | | | | | | | X |
| Serum chemistry (20-panel) <sup>f</sup> | X | | | | | | | | | X |
| Serum calcium (local)** | X | X | | | | | | | | |
| Serum calcium, phosphate, and albumin | X | | X | X | X | X | X | X | X | X |
| Serum calcium, potassium, sodium <sup>g</sup> | | | | | X | X | X | X | X | X |
| Serum 25-hydroxyvitamin D | X | | X | X | X | X | X | X | X | X |
| Serum 1,25-dihydroxyvitamin D | | | | | | X | | | | X |
| Serum bone turnover markers | X | | | X | X | X | | X | | X |
| Serum thyroid function test <sup>f,h</sup> | X | | | | | | | | | |
| Creatinine clearance (estimated GFR) | X | | | | X | | X | | | X |
| PTH and ECP antibodies <sup>i</sup> | X | | | | | X | | X | | $X^{l}$ |
| Serum PTH [1-84] for pharmacokinetic analysis | | | | | | | | | Xm | |
| FSH (newly menopausal women only) | X | | | | | | | | | |
| Serum pregnancy test (WOCBP only) | X | | | | X | X | X | X | X | X |
| Urine pregnancy test (WOCBP only) | X | | X | X | | | | | | |
| Urinalysis | X | | | | | | | | | X |
| 24-hour urine calcium, phosphate, sodium, creatinine | X | | | | X | | X | | | X |

Document: Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link

Author: 


| Visit Number | | Int. | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Procedures / Proposed Study Week <sup>a</sup> | | 1 <sup>c</sup> | 4 | 8 | 16 | 24 | 32 | 40 | 48 | 52 |
| Visit Windows | ± 3 days | ± 2 days | ± 7 days | ± 7<br>days | ±7 days | ± 7 days | ± 7 days | ± 7 days | ± 7 days | ± 7<br>days |
| Diary review <sup>j</sup> | | | X | X | X | X | X | X | X | X |
| Dispense/administration/accountability of study drug and pen injectors/ancillary supplies | X | | X | X | X | X | X | X | X | X |
| Dispense/accountability of calcium/calcitriol supplements (see guideline) | X | | X | X | X | X | X | X | X | X |
| Dispense subject diaries | X | | | | | | | | | X |
| Collect used/unused study drug and supplementsk | | | X | X | X | X | X | X | X | X |

 $BL = baseline; DXA = dual-energy \ x-ray \ absorptiometry; ECP = \textit{E.coli} \ protein; FSH = follicle \ stimulating \ hormone; GFR = glomerular \ filtration \ rate; Int. = interim \ visit;$ 

PTH = parathyroid hormone; WOCBP = women of child-bearing potential

Document: Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link

Author: 


<sup>\*</sup>Note: Final RELAY study parameters may be used as baseline parameters for this study.

<sup>\*\*</sup>Any adjustment of study drug or supplemental calcium and calcitriol doses requires testing of total serum calcium concentrations at interim time points.

<sup>&</sup>lt;sup>a</sup> Study visits will be conducted at Weeks 1 (baseline), 4, 8, every 8 weeks thereafter through Week 48, and at Weeks 52.

<sup>&</sup>lt;sup>b</sup> Week 8 from the RELAY study; subjects will return all used/unused drug, supplements, and pens from RELAY/REPLACE.

<sup>&</sup>lt;sup>c</sup> After the End of Treatment visit or early termination visit, subjects who will not continue rhPTH[1-84] treatment will have their total serum calcium and phosphate levels measured 3 to 5 days after the last dose of study medication. Doses of calcium and active vitamin D supplements will be adjusted by the Investigator as appropriate. Thereafter, the Investigator will repeat serum calcium/phosphate monitoring and supplement dose adjustments as appropriate to achieve target serum calcium/phosphate concentrations until the follow up phone call 4 weeks ± 7days after end of treatment visit. After the 4 week follow up phone call, further management of hypoparathyroidism will occur as part of the subject's long-term non-study medical care.

<sup>&</sup>lt;sup>d</sup> Vital signs should be done prior to blood draws.

<sup>&</sup>lt;sup>e</sup> Calcium supplements should be withheld for 24 hours prior to the DXA scan. If a subject cannot withhold the calcium supplements due to safety concern, the DXA should be performed 2 hours after the last calcium tablet has been ingested. Please note: DXA will NOT be completed at baseline if subject had a scan performed within the past 6 months in one of the previous studies (all subjects will have a DXA performed at Week 52 (Visit 9)

<sup>&</sup>lt;sup>f</sup> Fasting for at least 6 to 8 hours prior to test

g Serum potassium, sodium, and calcium is to be collected 1 week and again 1 month following the institution or change in dose of a calcium-sparing diuretic and then at each subsequent scheduled clinic visit.

h Thyroid function tests done for final visit of the RELAY/REPLACE studies only.

<sup>&</sup>lt;sup>i</sup> Blood draw for PTH and ECP antibodies will be done predose.

<sup>&</sup>lt;sup>1</sup> A paper diary will be dispensed at baseline for the investigator's use to assess subject's compliance and adherence to the protocol procedures.

<sup>&</sup>lt;sup>k</sup> Subject is to return unused and used cartridges and supplements at each visit.

<sup>&</sup>lt;sup>1</sup> See Protocol Section 6.2 for instructions on follow-up for subjects with PTH-specific antibodies and Table 6-3 for a schedule of follow-up procedures for these subjects.

m Blood samples for pharmacokinetic analysis will be drawn predose (0 hour) and postdose between 1 and 2 hours and between 6 and 10 hours following study drug administration.

Table 4. 2 Schedule of Evaluations and Procedures – Long-term Extension to Month 36

| Study Procedures / Proposed Study Month <sup>a, b</sup> | Months 14/26 | Months 16/28 | Months 18/30 | Months 20/32 | <b>Months 22/34</b> | Months 24/36** |
|---|---|---|---|---|---|---|
| Visit Windows | ± 2 weeks | ± 2 weeks | ± 2 weeks | ± 2 weeks | ± 2 weeks | ± 2 weeks |
| Concomitant medications | X | X | X | X | X | X |
| Adverse event monitoring, including pen-related events/complaints | X | X | X | X | X | X |
| Assessment of clinical episodes of hypocalcemia and hypercalcemia | X | X | X | X | X | X |
| Physical examination | | | X <sup>c</sup> | | | X <sup>c</sup> |
| Vital signs <sup>d</sup> and weight | X | X | X | X | X | X |
| Bone mineral density by DXA <sup>e</sup> | | | | | | X <sup>f</sup> |
| Hematology <sup>g</sup> | | | | | | X |
| Serum chemistry (20-panel) <sup>g</sup> | | | | | | X |
| Serum calcium (local)* | | | | | | |
| Serum calcium, phosphate | X | X | X | X | X | X |
| Serum calcium, potassium, sodium <sup>h</sup> | X | X | X | X | X | X |
| Serum 25-hydroxyvitamin D | X | X | X | X | X | X |
| Serum 1,25-dihydroxyvitamin D | | | X | | | X |
| Serum bone turnover markers | | X | | X | | X |
| Creatinine clearance (estimated GFR) | | X | | X | | X |
| PTH and ECP antibodies <sup>i, j</sup> | | | X | | | X |
| Serum pregnancy test (WOCBP only) | | | | | | |
| Urine pregnancy test (WOCBP) | X | X | X | X | X | X |
| Urinalysis | | | | | | |
| 24-hour urine calcium, phosphate, sodium, creatinine | | X | | X | | X |
| Diary review <sup>k</sup> | X | X | X | X | X | X |
| Dispense/administration/accountability of study drug, calcium, and pen injectors/ancillary supplies | X | X | X | X | X | X |
| Collect used/unused study drug and pen injectors <sup>1</sup> | X | X | X | X | X | X |

Document: Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link
Author: Version Numbers

Author: 


DXA = dual-energy x-ray absorptiometry; ECP = E. coli protein; EoT = end of treatment; F/up = follow up; GFR = glomerular filtration rate; Int.= interim visit; PTH = parathyroid hormone; WOCBP = women of child-bearing potential)

- <sup>a</sup> Study visits will be conducted every 2 months during the extension portion and will continue until the subject voluntarily withdraws or until termination of the study.
- b After the End of Treatment visit or early termination visit, subjects who will not continue rhPTH[1-84] treatment will have their total serum calcium and phosphate levels measured 3 to 5 days after the last dose of study medication. Doses of calcium and active vitamin D supplements will be adjusted by the Investigator as appropriate. Thereafter, the Investigator will repeat serum calcium/phosphate monitoring and supplement dose adjustments as appropriate to achieve target serum calcium/phosphate concentrations until the follow up phone call 4 weeks ± 7days after end of treatment visit. After the 4 week follow up phone call, further management of hypoparathyroidism will occur as part of the subject's long-term non-study medical care.
- <sup>c</sup> Brief physical exams will be conducted at 6-month intervals.
- <sup>d</sup> Vital signs should be done prior to blood draws.
- <sup>c</sup> Calcium supplements should be withheld for 24 hours prior to the DXA scan. If a subject cannot withhold the calcium supplements due to safety concern, the DXA should be performed 2 hours after the last calcium tablet has been ingested.
- f DXA will be performed at End of Treatment visit ONLY if the previous DXA was ≥3 months prior.
- g Fasting for at least 6 to 8 hours prior to test
- h Serum potassium, sodium, and calcium is to be collected 1 week and again 1 month following the institution or change in dose of a calcium-sparing diuretic and then at each subsequent scheduled clinic visit.
- <sup>1</sup> Blood draw for PTH and ECP antibodies will be done predose.
- <sup>j</sup> See Protocol Section 6.4.9 for instructions on follow-up for subjects with PTH-specific antibodies and Table 6-4 for a schedule of follow-up procedures for these subjects.
- k Subjects will record diary information during the 2-week period prior to the next scheduled visit during the long-term extension portion of the study. If the subject does not record the diary information as indicated during this time period, he/she may record it during the 2 weeks following the visit, for review at the next visit or via phone.
- <sup>1</sup> Subjects are to return unused and used cartridges at each visit. Pens will be collected at the final visit.

Document: Author: 

PPD

2.0

<sup>\*</sup>Any adjustment of study drug or oral calcium and active vitamin D doses requires testing of total serum calcium concentrations at interim time points.

<sup>\*\*</sup>Following Month 24, the every 2-month visit schedule will repeat (ie, visits procedures for Month 26 are the same as those shown at Month 14.)

Table 4. 3 Schedule of Evaluations and Procedures – Long-term Extension after Month 36

| Proposed Study Month <sup>a</sup><br>Study Procedures | Months 38/50/62 | Months 40/52/64 | Months 42/54/66 | Months 44/56/68 | Months 46/58/70 | Months 48/60/72 | End of<br>Treatment <sup>b</sup> | 4 weeks<br>F/up<br>Phone <sup>c</sup> |
|---|---|---|---|---|---|---|---|---|
| Visit Windows | ± 2 weeks | ± 2 weeks | ± 2 weeks | ± 2 weeks | ± 2 weeks | ± 2 weeks | ± 1 week | ±7 days |
| Re-consent subject <sup>d</sup> | X | | | | | | | |
| Concomitant medications | X | X | X | X | X | X | X | |
| Adverse event monitoring, including pen-related events/complaints | X | X | X | X | X | X | X | X |
| Assessment of clinical episodes of hypocalcemia and hypercalcemia | X | X | X | X | X | X | X | |
| Physical examination <sup>e</sup> | | | Xe | | | X <sup>d</sup> | X | |
| Vital signs <sup>f</sup> and weight | X | X | X | X | X | X | X | |
| Electrocardiogram (12-lead) | | | | | | | Xg | |
| Bone mineral density by DXAh | | | | | | X | Xi | |
| Hematology <sup>j</sup> | | | | | | X | X | |
| Serum chemistry (20-panel) <sup>j</sup> | | | | | | X | X | |
| Serum calcium (local)* | | | | | | | | |
| Serum calcium, phosphate | X | X | X | X | X | X | X | |
| Serum calcium, potassium, sodium <sup>k</sup> | X | X | X | X | X | X | X | |
| Serum 25-hydroxyvitamin D | X | X | X | X | X | X | X | |
| Serum 1,25-dihydroxyvitamin D | | | X | | | X | X | |
| Serum bone turnover markers | | X | | X | | X | X | |
| Creatinine clearance (estimated GFR) | | X | | X | | X | X | |
| PTH and ECP antibodies <sup>1</sup> | | | X | | | X | X <sup>m</sup> | |
| Serum pregnancy test (WOCBP only) | | | | | | | X | |
| Urine pregnancy test (WOCBP) | X | X | X | X | X | X | | |
| Urinalysis | | | | | | | X | |
| 24-hour urine calcium, phosphate, sodium, creatinine | | X | | X | | X | X | |
| Diary review <sup>n</sup> | X | X | X | X | X | X | X | |
| Dispense/administration/accountability of study drug, and pen injectors/ancillary supplies <sup>o</sup> | X | X | X | X | X | X | X | |
| Collect used/unused study drug / pen injectors <sup>p</sup> | X | X | X | X | X | X | X | |

Document: Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link
Author: Version Number:

Author: 


| Study Procedures | Proposed Study Month <sup>a</sup> | Months 38/50/62 | Months<br>40/52/64 | Months 42/54/66 | Months<br>44/56/68 | Months<br>46/58/70 | Months 48/60/72 | End of<br>Treatment <sup>b</sup> | 4 weeks<br>F/up<br>Phone <sup>c</sup> |
|---|---|---|---|---|---|---|---|---|---|
| | Visit Windows | ± 2 weeks | ± 2 weeks | ± 2 weeks | ± 2 weeks | ± 2 weeks | ± 2 weeks | ± 1 week | ± 7 days |

DXA = dual-energy x-ray absorptiometry; ECP = *E. coli* protein; EoT = end of treatment; F/up = follow up; GFR = glomerular filtration rate; Int.= interim visit; PTH = parathyroid hormone; WOCBP = women of child-bearing potential

NOTE: Following Month 72, the every 2-month visit schedule will repeat (ie, visits procedures for Month 74 will repeat starting with those shown at Months 26/38/50.)

- \*Any adjustment of study drug or oral calcium and active vitamin D doses requires testing of total serum calcium concentrations at interim time points.
- <sup>a</sup> Study visits will be conducted every 2 months and will continue until the subject voluntarily withdraws or until termination of the study (**currently extended at least until December 2016**). At that time, and periodically following the December 2016 milestone, the study will be reviewed in regard to continuation/termination status.
- <sup>b</sup> After the End of Treatment visit or early termination visit, subjects who will not continue rhPTH[1-84] treatment will have their total serum calcium and phosphate levels measured 3 to 5 days after the last dose of study medication. Doses of calcium and active vitamin D supplements will be adjusted by the Investigator as appropriate. Thereafter, the Investigator will repeat serum calcium/phosphate monitoring and supplement dose adjustments as appropriate to achieve target serum calcium/phosphate concentrations until the follow up phone call 4 weeks ± 7days after end of treatment visit. After the 4 week follow up phone call, further management of hypoparathyroidism will occur as part of the subject's long-term non-study medical care.
- <sup>c</sup> Follow-up phone contact 4 weeks after the last dose of study medication to check on any ongoing or new drug-related AEs or SAEs
- <sup>d</sup> Study subjects must be re-consented at their next study visit prior to implementation of Amendment 5.
- <sup>e</sup> Brief physical exams will be conducted at 6-month intervals.
- f Vital signs should be done prior to blood draws.
- g The End of Treatment ECG will be read locally.
- h Calcium supplements should be withheld for 24 hours prior to the DXA scan. If a subject cannot withhold the calcium supplements due to safety concern, the DXA should be performed 2 hours after the last calcium tablet has been ingested.
- <sup>i</sup> DXA will be performed at End of Treatment visit ONLY if the previous DXA was ≥3 months prior.
- <sup>j</sup> Fasting for at least 6 to 8 hours prior to test
- k Serum potassium, sodium, and calcium is to be collected 1 week and again 1 month following the institution or change in dose of a calcium-sparing diuretic and then at each subsequent scheduled clinic visit.
- <sup>1</sup> Blood draw for PTH and ECP antibodies will be done predose.
- m See Protocol Section 6.4.9 for instructions on follow-up for subjects with PTH-specific antibodies and Table 6-4 for a schedule of follow-up procedures for these subjects.
- <sup>n</sup> Subjects will record diary information during the 2-week period prior to the next scheduled visit during the long-term extension portion of the study. If the subject does not record the diary information as indicated during this time period, he/she may record it during the 2 weeks following the visit, for review at the next visit or via phone.
- <sup>o</sup> Ancillary supplies (ie, needles and alcohol wipes) may be supplied, as allowed by local regulations.
- <sup>p</sup> Subjects are to return unused and used pen injectors at each visit.

Document: Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link

Author: 


Table 4. 4 Schedule of Follow-up Visits and Procedures for Subjects with PTH-specific Antibodies at Final Visit

| Follow-up Procedures <sup>a</sup> | Follow-up<br>(Month 3)b | Follow-up<br>(Month 6) |
|---|---|---|
| Visit Number: | F3 | F4 |
| Visit Window (± Days) | ±7 | ±7 |
| Antibodies to PTH | X | X |
| Adverse events | X | X |

AE = adverse event; F = follow-up; PTH = parathyroid hormone

Document: Author:  Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link
PPD Version Number

Version Number: Version Date: 2.0

sion Date: March 22, 2018

<sup>&</sup>lt;sup>a</sup> Follow-up visits will be conducted for only those subjects who are determined to have PTH-specific antibodies at the end of the End of Study visit (or at the time of discontinuation) and are NOT continuing treatment on commercial Natpara.

<sup>&</sup>lt;sup>b</sup> Subjects who have negative antibody results at Month 3 do not need the Month 6 follow-up visit.

#### 4.2. **Efficacy Endpoint**

The proportion of subjects in whom the following three conditions are fulfilled at Week 52 (Visit 9) and/or at the End of Treatment will be summarized:

- $A \ge 50\%$  reduction from baseline in dose of oral calcium supplementation or an oral calcium dose of  $\leq 500 \text{ mg AND}$
- $A \ge 50\%$  reduction from baseline in dose of oral calcitriol supplementation or an oral calcitriol dose of  $\leq 0.25 \mu g$  AND
- An albumin-corrected total serum calcium concentration that is normalized or maintained compared to the baseline value and does not exceed the ULN for the central laboratory

#### 4.3. **Other Efficacy Endpoints**

- Mean percentage changes from baseline in supplemental oral calcium and supplemental calcitriol dosages at each visit
- Proportion of subjects achieving the three conditions of the efficacy endpoint defined above at each visit
- Mean change from baseline in 24-hour urine calcium excretion
- Impact of calcium source (carbonate vs. citrate) on response
- Impact of calcium-sparing diuretics on serum and urinary calcium
- Proportion of subjects that maintain a calcium phosphate product in the range of 35 to  $55 \text{ mg}^2/dL^2$
- Distribution of subjects by rhPTH[1-84] doses at the End of Treatment Visit
- Change from baseline in bone turnover markers, bone-specific alkaline phosphatase, serum carboxy-terminal telopeptide of type I collagen, serum procollagen type 1 aminoterminal propeptide, osteocalcin, PTH antibodies, and BMD by DXA
- Additional subgroup analyses that are specified in the SAP

#### 4.4. **Exploratory Endpoints**

There is no exploratory endpoint specified for this study.

#### 4.5. **Safety Endpoints**

The safety endpoints include:

- Adverse events and serious adverse events
- Incidence of adverse events of hypocalcemia (eg, paresthesia, numbness, tetany) and hypercalcemia (eg, constipation, nausea, poor appetite or vomiting, frequent urination, thirst, and kidney stones)
- Incidence of hypercalciuria
- Laboratory test results

PPD

o Hematology (hematocrit, hemoglobin, white blood cells, red blood cells, platelets, differential)

Document: Author:

- o Serum chemistries (standard Chem-20 panel, including calcium, phosphorus, and albumin)
- Serum 25-hydroxyvitamin D levels
- Serum 1,25-dihydroxyvitamin D levels
- Creatinine clearance
- o Serum bone turnover markers
- o Urinalysis
- o 24-hour urine calcium, phosphate, sodium, and creatinine excretion
- o PTH and E. coli protein (ECP) antibodies
- Bone mineral density (BMD) by dual-energy x-ray absorptiometry (DXA)
- Electrocardiogram (ECG) parameters
- Physical examinations (including vital signs)
- Reason for termination from the study

Document: Author:

#### 5. **Statistical Methods**

#### 5.1. **General Methodology**

All statistical procedures will be completed using SAS version 9.4<sup>1</sup>. No formal statistical testing will be conducted for this study. Summary statistics will be provided.

Continuous variables, including those assessed on a discrete scale, will be summarized using descriptive statistics including number of subjects, mean, median, standard deviation, maximum, and minimum. For categorical variables, statistical summaries will include number of subjects and percentages.

For summary purposes, baseline will be defined as the last available pre-dose value, unless otherwise specified. End of treatment (EOT) time point, defined as the last determination of response or last available measurement during the treatment period (from the date of first dose to the date of last dose + 1 day), will be analyzed in addition to the scheduled visits. Visits will be summarized based on the analysis visit windows.

#### 5.2. **Adjustments for Covariates**

No preselected covariates are selected for adjustments.

#### 5.3. **Visit Windows**

#### 5.3.1. **Analysis Visit Windows**

Analysis visit windows are defined in Table 4.

Table 5. 1 Analysis Visit Window Definition (1st 12 Month of Study)

| Analysis Visit | Target Study Day | Analysis Visit Window |
|---|---|---|
| Baseline | 1 | See definition in Section 7.3.2 |
| Week 4 | 29 | [2, 42], and ≤last dose day + 1 |
| Week 8 | 57 | [43, 84], and ≤last dose day + 1 |
| Week 16 | 113 | [85, 140], and ≤last dose day + 1 |
| Week 24 | 169 | [141, 196], and ≤last dose day + 1 |
| Week 32 | 225 | [197, 252], and ≤last dose day + 1 |
| Week 40 | 281 | [253, 308], and ≤last dose day + 1 |
| Week 48 | 337 | [309, 350], and ≤last dose day + 1 |
| Week 52 | 365 | ≥351, and ≤last dose day + 1 or <start date="" extension="" of="" period<="" td="" the=""></start> |

If there are more than one non-missing observations in the same analysis visit window, the following selection rules will be applied sequentially to determine which observation will be used for analysis:

- The observation that is closer to the target day will be used;
- If Observations are equal-distance in days from the target day, the later one based on measurement date and time will be used.

Document: Author:

PPD

Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link

Version Number:

2.0


Analysis visit in the Long Term Extension period will be the same as the nominal visit in the CRF database. No derivation is necessary.

#### 5.3.2. **Definition of Baseline**

For all data including baseline variables, efficacy endpoints, and safety endpoints, the baseline values are defined as follow:

- For subjects who previously completed the REPLACE and RELAY studies or completed only the REPLACE study, the baseline value of REPLACE study will be used as the baseline value for this study;
- For subjects who previously only completed RELAY study, the baseline value of RELAY study will be used as the baseline value for this study;
- For subjects who enrolled in REPLACE and dropped out during optimization and subjects who are new to the rhPTH[1-84] treatment, Visit 1 (BL visit) record of this study will be used as the baseline value.

#### 5.4. Handling of Dropouts or Missing Data

#### 5.4.1. Handling of Dropouts or Missing Data for Efficacy Analysis

The daily dose of calcium and vitamin D metabolite/analog will be computed based on both investigator prescribed data and subject diary data. The investigator prescribed data will be considered as the primary method for all efficacy analysis endpoints.

The daily dose of calcium and vitamin D metabolite/analog based on investigator prescription will be determined by using the latest prescribed dose prior to the assessment date of albumin corrected calcium for each analysis visit. To avoid the effect of potential fluctuation of the supplemental medication dose, the prescribed supplemental medication dose at Visit 1 (BL visit) will be excluded from the derivation of the baseline dose and the prescribed dose at the Visit 9 (week 52) for subjects who complete the treatment or Early Termination Visit. Subjects that discontinued early will be excluded from the derivation of the post-baseline prescribed dose.

The average daily dose of calcium and vitamin D metabolite/analog based on subject diaries will be calculated as the average daily dose of a 14-day interval. The 14-day interval for each current analysis visit includes the dose reported during the 14 days on or prior to the assessment date of albumin corrected calcium. However, this 14-day interval should not include or go beyond the assessment date of albumin corrected calcium for the previous analysis visit. If the number of days from the previous albumin corrected calcium date to the current assessment date is less than 14 days, the actual number of days during the two analysis visits will be used to calculate the average daily dose. If the number of days from the previous albumin corrected calcium date to the current assessment date is less than 9 days, the average daily dose will not be calculated and will be classified as missing. Diary data after the last dose date of study drug will be excluded from the derivation.

A missing daily dose of calcium and vitamin D from subject diaries will not be imputed. A minimum 9 days of non-missing data from the intervals is required, otherwise the average daily dose will be classified as missing. Because recordings of dose of calcium and vitamin D metabolite/analog may be missing on different days, different days within the interval may be used in the computation for the daily dose of calcium and for the daily dose of vitamin D metabolite/analog.

For determination of baseline supplemental medication dose, the derivation rules specified in this section will only be applicable when the value of Visit 1 (BL visit) of this study is used as the baseline value. For all other cases, as specified in section 7.3.2, baseline values will be obtained from the REPLACE or RELAY study. The detailed derivation rules are provided in the SAPs for REPLACE and RELAY studies accordingly.

Document: Author:

PPD

#### 5.4.2. Handling of Dropouts or Missing Data for Safety Analysis

Missing safety parameters will not be imputed.

#### 5.4.3. **Handling of Partial Dates**

Complete dates will be imputed from partial dates of adverse events and medications solely for the purpose of defining treatment emergence for adverse events and prior/concomitant status for medications. Dates will be defined using the hierarchy of derivations below.

Adverse event or medication start date:

- 1. If year and month are known, and it is the month and year of the first dose date, use the first dose date.
- 2. If year and month are known, and it is the month and year of the informed consent, use the informed consent date.
- 3. If year and month are known, and the month is not the month and year of the first dose or informed consent, use the first day of the month.
- 4. If only year is known, and it is previous to the year of the informed consent, use June 30<sup>th</sup> of that year.
- 5. If only year is known, and it is the year of the informed consent, use the informed consent date.
- 6. Should any of the previous start dates created be after a complete stop date provided, use the stop date instead of the date that would otherwise be created.
- 7. Otherwise, if start date is unknown leave as missing.

## Medication stop date:

- 1. If year and month are known and study medication stopped during that month and year, use the stop date of study medication.
- 2. If year and month are known and informed consent was provided during that month and year, use the date of informed consent.
- 3. If year and month are known and study medication stopped after the date of informed consent and not in the month that medication stopped, use the last day of the month.
- 4. If year and month are known and are prior to the month of informed consent, use the first day of the month.
- 5. If only year is known and study medication stopped during that year, use the stop date of study medication.
- 6. If only year is known and study medication stopped after that year, use December 31st of that year.
- 7. If only year is known and study medication stopped prior to that year, use the first day of the year.
- 8. Should any of the previous stop dates created be before a start date, either a complete date or an imputed one, use the (imputed) start date instead of the date that would otherwise be created.
- 9. Otherwise, if stop date is unknown leave as missing.

#### 5.5. **Interim Analyses and Data Monitoring**

Two interim study reports will be completed: 3-year interim analyses to look at safety and efficacy compiled through 31 May, 2013; 5-year interim analyses to look at safety and efficacy compiled through 08 May 2017. There is no DSMB identified for this study.

#### 5.6. **Multicenter Studies**

Center will not be used as a covariate factor in the analysis.

## 5.7. Multiple Comparisons/Multiplicity

Not applicable.

## 5.8. Active-Control Studies Intended to Show Non-inferiority or Equivalence

There is no active control in the current study

## 5.9. Examination of Subgroups

Subgroup analysis by gender will be performed for the primary efficacy endpoint. Additional subgroup analysis may be explored as appropriate. Subgroup results need to be interpreted with caution if there is insufficient number of subjects in a subgroup.

Document: Author:  Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link PPD Version Number:


2.0

#### 6. **Statistical Analysis**

#### 6.1. **Disposition of Subjects**

Subject disposition will be summarized for all subjects enrolled as well as subjects in each analysis population.

The number and percentage of subjects assessed at each planned visit, subjects completing the treatment (based on the study exit CRF at Visit 9 (week 52), completing the study (based on the study exit CRF and finish the follow-up Visit 11 (week 56), and discontinuation by reasons will be summarized

#### 6.2. **Protocol Deviations**

Protocol deviations will be identified programmatically as well as based on protocol deviations collected by the study monitors. A summary table and listing of all collected protocol deviations might be presented upon request.

#### 6.3. **Analysis Populations**

The analysis populations to be used in this study are the Safety Population and the Intent-to-Treat (ITT) Population.

The Safety Population includes all subjects who received at least one dose of study drug with any follow-up information. All safety analyses will be conducted on this population.

The ITT population includes all subjects who received at least one dose of study drug and had at least one efficacy measurement. The primary and secondary efficacy analyses will be based on the ITT population.

#### 6.4. **Demographic and Other Baseline Characteristics**

Demographic variables (such as sex, age, race, etc.) and medical history will be obtained; medical history will be reviewed and updated as necessary from the RELAY or REPLACE study, if available, for subjects previously enrolled in those studies.

Descriptive statistics will be used to summarize the baseline and demographic characteristics. Demographic and baseline characteristics to be presented include:

- age (in years, both as a continuous parameter and by categories of <45, 45-64, >=65)
- gender
- race •
- ethnicity
- height (cm) at the baseline visit
- weight (kg) at the baseline visit
- body mass index (BMI) (kg/m<sup>2</sup>) at the baseline visit

Medical and surgical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA)<sup>2</sup>, Version 13.0. The history will be summarized by system organ class (SOC) and preferred term (PT) within system organ class for the Safety Population, with both SOC and PT sorted alphabetically.

#### 6.5. **Measurements of Treatment Compliance**

The data for study medication use are reported in the paper diary. Percent treatment compliance will be calculated as:

[100\*doses administered / days on treatment], where days on treatment is calculated as (date of last dose - date of first dose) + 1.

Document: Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link Subjects will be considered compliant overall for study medication if the calculated compliance is ≥80% to ≤120%. Overall treatment compliance will be presented using descriptive statistics and the number and percentage of subjects who are ≥80% to ≤120% compliant will be presented for the Safety Population.

#### 6.6. **Extent of Exposure**

#### 6.6.1. **Exposure during this (RACE) study**

The extent of exposure is defined as the number of days on treatment, calculated as: (date of last dose - date of first dose) + 1.

The date of the first dose is based on CRF entry. The date of the last dose will be based on information collected in the paper diary. The extent of exposure and the number of days that the dose was administered will be summarized. The extent of exposure will also be categorized into weeks (<1, 1-<4, 4-<8, 8-<16, 16-<24, 24-<32, 32-<40, 40-<48, 48-<52, ≥52) and tabulated. Exposure summaries will be presented for the Safety Population. Number of subjects at different dose level at EOT will be summarized as specified in section 8.7.2.

#### 6.7. **Analysis of Efficacy**

All efficacy analyses will be conducted on the ITT Population.

Prescriptive analyses will be presented by visit in order to see how the status or value changes over time. The EOT status or value will be included as a separate time point in the summary.

Efficacy endpoints based on the calcium and/or calcitriol supplement will be derived using both the investigator prescribed data and subject diary data. Computation of daily calcium and calcitriol dose is specified in Section 7.4.1. Analysis based on the investigator prescribed data will be primary. Analysis based on the subject diary data will be considered as supportive.

#### 6.7.1. **Primary Analysis**

As specified in the definition of efficacy endpoint, the subject must meet three conditions at Week 52 and/or EOT to be considered a responder. First, the subject's prescribed daily oral calcium supplementation should be reduced by at least 50% from baseline or an oral calcium dose of  $\leq$  500 mg; second, the subject's prescribed daily oral calcitriol supplementation dose should be reduced by at least 50% from baseline or an oral calcitriol dose of  $\leq 0.25 \,\mu g$ . For the third condition, albumin-corrected total serum calcium concentration should be normalized or maintained compared to the baseline value (≥7.5 mg/dL) and does not exceed the ULN for the central laboratory. Different maintenance ranges for this third condition will be assessed in the sensitivity analysis (Section 8.7.5).

The calculation of daily calcium and calcitriol dose is specified in Section 7.4.1. The determination of responders using the subject diary dose data instead of prescribed dose will be used as one of the supportive analyses to the primary analysis.

The number and percentage of responder status will be presented. No formal statistical test will be done. A bar chart for percent of subjects who achieve responder status will be plotted. The percent of subjects who achieve calcium supplement response criterion, and the percent of subjects who achieve calcitriol supplement response criterion will also be plotted in a bar chart.

No statistical testing will be conducted to compare between group differences.

## 6.7.2. Other Analyses

## Mean percentage changes from baseline in supplemental oral calcium and supplemental calcitriol dosage at each visit

The absolute and percentage changes from baseline will be summarized at each visit. No formal statistical test will be done.

## Proportion of subjects achieving the primary endpoint at each visit

The number and percentage of subjects achieving the primary efficacy endpoint will be presented by visit. No formal statistical test will be done.

## Mean percentage change from baseline in 24-hour urine calcium excretion

The absolute and percentage changes from baseline will be summarized by visit. No formal statistical test will be done.

## Impact of calcium source (carbonate vs. citrate) on response

The number and percentage of subjects meeting the criteria of being responders will be presented by visit and by calcium source (carbonate vs. citrate). No formal statistical test will be done.

## Impact of calcium-sparing diuretics on serum and urinary calcium

The number and percentage of subjects who use at least one calcium-sparing diuretics during the study will be presented.

The urinary calcium will be listed for subjects who received calcium-sparing diuretics during the study. No formal statistical test will be done.

# <u>Proportion of subjects that maintain a calcium phosphate product in the range of 35 to 55</u> $mg^2/dL^2$

Calcium phosphate product will be classified as normal (35 - 55 mg²/dL²), or abnormal (including low and high). The number and percentage of subjects with maintenance of a calcium phosphate product in the normal range will be presented by visit. No formal statistical test will be done.

## Distribution of subjects by rhPTH[1-84] doses at the End of Treatment Visit

The number and percentage of subjects at different dose levels at the EOT visit will be summarized. No formal statistical test will be done.

# Change from baseline in bone turnover markers (bone-specific alkaline phosphatase, serum carboxy-terminal telopeptide of type I collagen, serum procollagen type 1 amino-terminal propeptide, and osteocalcin), PTH and ECP antibodies, and BMD by DXA

The absolute and percentage changes from baseline will be summarized by visit. No formal statistical test will be done. For DEXA, Z-scores will also be presented and summarized.

## 6.7.3. Subset Analyses

Subgroup analyses will be done as specified in Section 7.9.

## 6.7.4. Exploratory Analyses

There is no exploratory analysis planned.

Document:
Author:


Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link
Version Number:
Version Date:
March 22, 2018

## 6.7.5. Sensitivity Analyses

There is no sensitivity analysis planned for this study.

## 6.8. Analysis of Safety

All safety analyses will be performed on the Safety Population. All values presented in summaries will be observed values. No formal statistical comparisons are planned.

### **6.8.1.** Adverse Events

Adverse events will be coded using MedDRA Version 13.0. Adverse event listings will provide the verbatim term as well as SOC and PT for each recorded event. A separate listing may be produced to provide the SOC, high level term, PT, and lower level term that are associated with each verbatim term.

Treatment emergent adverse events (TEAEs) are defined as AEs whose onset occurs, severity worsens or intensity increases after receiving the study medication of this study and <= 30 days after last dose of study drug. If any AE records contain only partial dates, these will be handled by imputation, as described in Section 7.4.3. AEs which are not treatment emergent will be flagged in listings.

An overview of TEAEs will be summarized using the number and percentage of subjects. The number of events will also be presented except for summaries by highest category. Categories summarized will include any TEAEs, severity of TEAEs (any and highest category), relationship of TEAEs to treatment (any and highest category), treatment emergent serious AEs (TESAEs), severity of TESAEs, relationship of TESAEs to treatment, TEAEs leading to discontinuation, and TEAEs leading to death.

Treatment emergent AEs will be summarized using number and percentage of subjects. Subject incidence for AEs within each SOC and PT will be presented, and the number of events will also be summarized except for summaries by highest category. Categories summarized will be the same as those summarized overall, except that no summary table will be provided for TEAEs leading to death.

Summaries of TEAEs and TESAEs will also be presented by PT. These presentations will be sorted by descending incidence.

Listings will be provided for serious adverse events (SAEs), AEs leading to discontinuation, and AEs leading to deaths.

The incidence of hypocalcemia and hypercalcemia will be identified by clinical preview. Prevalence of hypocalcemia and hypercalcemia will be assessed at all visits on the date of visit. The number of subjects with hypocalcemia and hypercalcemia and the number of episodes of hypocalcemia and hypercalcemia will be assessed for the overall trial.

## 6.8.2. Clinical Laboratory Evaluation

All laboratory parameters will be collected and processed via a central laboratory, with exception of all urine pregnancy tests and total serum calcium levels which will be done at investigator's local laboratories. Standard international (SI) units will be used for data presentation. Only scheduled lab parameters will be included in the lab summaries. All lab data will be included in the listings.

Quantitative results will be summarized for hematology, serum chemistry, thyroid function tests (levothyroxine and thyroid-stimulating hormone), creatinine clearance, urinary chemistries (24-hour urine calcium, phosphate, and sodium excretion), and selected urinalysis parameters (pH, specific gravity, and urobilinogen) by visit. Both actual values and change from baseline will be summarized. Additionally, shift tables will be presented, summarizing cross tabulations of low,

Document: Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link Author: Version Number

Version Number: 2.0 Version Date: March 22, 2018 normal, and high based on the parameter normal range, from baseline to each post-baseline visit and EOT. Percentages for shift tables will be based on the number of subjects with both baseline and post-baseline values at each visit.

Categorical urinalysis findings and urine pregnancy results will be presented in appendix data listings only.

Estimated creatinine clearance rate will be re-calculated based on the Cockcroft-Gault (C-G) equation:

CLcr (mL/min) =  $[140 - age (years)] \times weight (kg) {\times 0.85 \text{ for female subjects}} / (72 \times serum creatinine (mg/dL)),$ 

Estimated creatinine clearance rate will be summarized by stages as defined in Table 5.

Table 6. 1 Definition of the Stages of Clcr3

| Stage | Description | CLcr (mL/min) |
|---|---|---|
| 1 | Control (normal) Glomerular filtration rate (GFR) | ≥ 90 |
| 2 | Mild decrease in GFR | 60-89 |
| 3 | Moderate decrease in GFR | 30-59 |
| 4 | Severe decrease in GFR | 15-29 |
| 5 | End Stage Renal Disease (ESRD) | <15 not on dialysis |
| | | Requiring dialysis |

The number and percentage of subjects with post-baseline results qualifying as markedly abnormal will be summarized by parameter. A listing of all values for the parameter which qualifies as markedly abnormal will be provided. Markedly abnormal laboratory criteria are defined in Table 6.

Table 6. 2 Markedly Abnormal Laboratory Criteria<sup>4</sup>

| Lab parameter | Unit | Lower Limit | Upper Limit |
|----------------------|--------|-------------|-------------|
| Chemistry | | | |
| Albumin | g/L | <=20 | >=90 |
| Alkaline Phosphatase | U/L | NA | >2*ULN |
| ALT | U/L | NA | >3*ULN |
| Amylase | U/L | <=15 | >=350 |
| AST | U/L | NA | >3*ULN |
| Bilirubin | μmol/L | NA | >2*ULN |
| BUN | mmol/L | NA | >=10.7 |
| Calcium (total) | mmol/L | <=2.1 | >=3.0 |
| Chloride | mmol/L | <=80 | >=125 |
| Cholesterol (total) | mmol/L | NA | >=12.9 |
| Creatinine | μmol/L | NA | >=177 |
| Creatinine clearance | ml/min | <=60 | NA |

Document: Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link

Author: 

Version Number: 2.0 Version Date: March 22, 2018

| Glucose | mmol/L | <=1.7 | >=13.9 |
|---|---|---|---|
| Gamma glutamyl transferase | U/L | NA | >=100 |
| Phosphate | mmol/L | NA | >=2 |
| Potassium | mmol/L | <=2.5 | >=6.5 |
| Sodium | mmol/L | <=120 | >=165 |
| Triglycerides | mmol/L | NA | >=5.6 |
| Uric acid | μmol/L | NA | >=624 (males)<br>>=505 (females) |
| | He | ematology | |
| Hematocrit | L/L | <=0.37 (males)<br><=0.32 (females) | >0.54 (males)<br>NA (females) |
| Hemoglobin | g/L | <=115 (males)<br><=95 (females) | NA |
| Platelets | $10^{9}/L$ | <=75 | >=700 |
| RBC count | $10^{12}/L$ | <=2.5 (males)<br><=2.0 (females) | NA |
| WBC count | 10 <sup>9</sup> /L | <=2.8 | >=16.0 |
| Basophils | L/L | NA | >=0.15 |
| Eosinophils | L/L | NA | >=0.10 |
| Lymphocytes | L/L | NA | >=0.80 |
| Monocytes | L/L | NA | >=0.40 |
| Neutrophils | L/L | <=0.15 | NA |
| - | 24- | Hour urine | |
| Urine calcium | mg | NA | >300 for men<br>>250 for women |

NA=Not Applicable; ULN = Upper Limit of Normal

## 6.8.3. ECG Evaluations

The number and percentage of subjects with each type of ECG finding (Normal/Abnormal, Not Clinically Significant/Abnormal, and Clinically Significant) will be presented by visit.

Actual value and change from baseline for each ECG parameters (HR, PR, QRS, QT, QTcB, QTcF) will be presented by visit.

Potentially clinically significant QTc finding criteria are defined in Table 7. The number and percentage of subjects with post-baseline results qualifying as potentially significant will be summarized by parameter. A listing will present all values for a subject and parameter for cases where at least one value for that parameter was potentially significant.

Table 6. 3 Potentially Clinically Significant Post-Baseline ECG<sup>5,6</sup>

| ECG Parameter | Potentially Clinical Significant Criterion |
|---------------|-----------------------------------------------------------|
| QTcB | ≥ 500 ms |
| QTcF | ≥ 500 ms |
| QTcB | An increase from Baseline of $\geq$ 60 ms or $\geq$ 30 ms |
| QTcF | An increase from Baseline of $\geq$ 60 ms or $\geq$ 30 ms |

## 6.8.4. Vital Signs, Physical Findings, and Other Observations Related to Safety

In general, other by-visit safety findings will be analyzed and presented in a way similar to laboratory variables.

## 6.8.4.1. Vital Signs

Vital signs to be analyzed include sitting blood pressure, sitting heart rate, and body temperature.

Document:
Author:

Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link
Version Number:
Version Date:
March 22, 2018

Observed vital signs and changes from baseline will be summarized by visit.

The number and percentage of subjects with post-baseline results qualifying as markedly abnormal will be summarized by parameter. A listing will present all values for a subject and parameter for cases where at least one value for that parameter was markedly abnormal. Post-baseline markedly abnormal vital signs criteria are defined in Table 8.

Table 6. 4 Markedly Abnormal Post-Baseline Vital Signs<sup>7</sup>

| Vital Sign Parameter | Abnormally Low | Abnormally High |
|---|---|---|
| Systolic blood pressure | A decrease from Baseline of $\geq$ 20 to a | An increase from Baseline of $\geq$ |
| (mmHg) | value ≤ 90 | 20 to a value $\geq$ 180 |
| Diastolic blood pressure | A decrease from Baseline of $\geq$ 15 to a | An increase from Baseline of ≥ |
| (mmHg) | value ≤ 50 | 15 to a value $\geq$ 105 |
| Heart Rate (bpm) | A decrease from Baseline of $\geq$ 15 to a | An increase from Baseline of ≥ |
| | value ≤ 50 | 15 to a value $\geq$ 120 |
| Temperature (°C) | N/A | Value $\geq$ 38.3°C and $\geq$ 0.8°C |
| 18 18 | | increase from Baseline |

## 6.8.4.2. Body Weight

The observed values and changes from baseline for body weight and BMI will be summarized at each visit.

## 6.8.4.3. Serum 25-Hydroxyvitamin D and Serum 1,25-dihydroxyvitamin D

The observed value and change from baseline in serum vitamin D levels (Serum 25-hydroxyvitamin D and Serum 1,25 vitamin D) will be summarized descriptively by visit.

## 6.8.4.4. Physical Examination Findings

Physical examination results will be presented in appendix data listings only.

## 6.8.4.5. PTH and ECP Antibodies

The number and percentage of subjects classified as having antibodies to PTH and ECP at baseline, Visit 5 (Week 24), Visit 7 (Week 40), and EOT will be tabulated for each treatment group.

If any subject tests positive for PTH-specific antibodies at the final visit, they will have follow-up blood draws for PTH antibody analysis at Months 2, 3, and 6 post-study. If a subject's results are negative at 2 successive visits within this timeframe, follow-up may be terminated. If at the end of 6 months the subject is still determined to have PTH-specific antibodies, the investigator and the sponsor will determine if additional follow-up may be required. During this time, subjects also will be evaluated for AEs or SAEs related to immunogenicity, which will be collected in the Pharmacovigilance database.

Subjects may remain on study if they develop PTH-specific antibodies during the study, providing that there are no concurrent AEs related to immunogenicity.

The number and percentage of subjects classified as having antibodies to PTH during the follow up period will also be provided, if applicable.

## 6.8.5. Concomitant Medications

Prior and concomitant medications will be coded to indication-specific ATC (Anatomic Therapeutic Chemical classification) and preferred name using the 1Q2010 version of the World Health Organization (WHO) Drug Dictionary.

Document: Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link
Author: Version Number


Version Number: 2.0 Version Date: March 22, 2018 Prior medications are defined as medications taken prior to the first dose of study medication in this study (RACE). Medications ongoing at the end of the previous study will be considered as prior medications. Concomitant medications are defined as medications that are taken during the treatment period of this study. Partial date imputation for medications is described in Section 7.4.3.

Prior and concomitant medication use will be summarized by level 2 ATC and preferred term using the number and percentage of subjects. Medications will be sorted alphabetically by ATC and preferred term within ATC. Subjects with multiple occurrences of a medication in ATC and preferred term will only be counted once within each ATC and preferred term. Since medications are coded to ATC by indication, preferred terms may appear under multiple ATCs.

#### 7. **Programming Conventions for Outputs**

Partial dates should be presented as --NOV1999 or ----- 1999 as needed.

Partial times should be presented as --: 30 or 14:-- as needed.

Listings should be sorted according to the order of the columns.

Document: Author:

Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link

Version Number: Version Date:

#### Mock Tables, Listings and Graphs (TLG) 8.

The mock TLGs will be provided in a separate document and will follow the numbering scheme described in ICH, E3, Guideline for Industry, "Structure and Content of Clinical Study Reports" for tables, subject data listings and graphs.

Document: Shire PAR-C10-008 SAP Amendment 1 v2.0 20180322 fix link PPD Author: Version Number:

#### 9. References

- 1. SAS Institute, Inc. SAS OnlineDoc Version Eight. SAS Institute, Inc, Cary, NC, 1999.
- 2. Medical Dictionary for Regulatory Activities (MedDRA), Version 13.0. IFPMA, International Committee on Harmonization. Geneva, Switzerland. 2010.
- 3. National Kidney Foundation. Clinical Practice Guidelines for Chronic Kidney Disease: Evaluation, Classification, and Stratification. Part 4, Definition and Stages of Chronic Kidney Disease. [Updated 2000].
- 4. Data on File. ACM Global Central Laboratory April 2010.
- 5. FDA Guidance Industry on E14 Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs, October 2005; 9-11.
- 6. Data on File. ERT Cardiac Solutions 2012.
- 7. Prohealthsys.com Canada: Bates Physical Assessment and Web MD [updated 2010].

Document: Author:


## Appendix I: Summary of Changes Made to SAP version 1.0 Dated October **10.** 24, 2011

Changes that are editorial in nature (to correct typographical errors, errors in formatting, or to modify the language) are not included.

| Section No. | SAP Version 1.0 | SAP Amendment 1 | Change Justification |
|---|---|---|---|
| Title | A <b>12-Month</b> Open-label Study | A Long Term Open-label<br>Study | In compliance to<br>Protocol Amendment 3,<br>Version 4.0 |
| Section 5.1 | | Add a bullet 'At the end of Week 52, subjects will be invited to extend their study drug regimen until at least October 2013. During this time, subjects will return to the clinic for interim visits every 2 months (Months 14, 16, 18, etc). | In compliance to<br>Protocol Amendment 3,<br>Version 4.0 |
| Section 5.1 | | Reordering of study visits to accommodate the long-term extension. | In compliance to<br>Protocol Amendment 3,<br>Version 4.0 |
| Section 5.1 | Figure 1 | Replaced by Figure 1.1 and Figure 1.2 | In compliance to<br>Protocol Amendment 3,<br>Version 4.0 |
| Section 5.3 | Approximately 40 subjects are anticipated to be enrolled. | Approximately 50 subjects are anticipated to be enrolled. | In compliance to<br>Protocol Amendment 3,<br>Version 4.0 |
| Section 6.1 | Table 1 Schedule of Study<br>Evaluations and Procedures | Replaced by Table 1, Table 2, and Table 3 | In compliance to<br>Protocol Amendment 3,<br>Version 4.0 |
| Section 6.1 | | Add lab assessments 'Serum 1,25-dihydroxyvitamin D levels' and ECP antibody | In compliance to<br>Protocol Amendment 3,<br>Version 4.0 |
| Section 6.2 | Section header: Primary<br>Efficacy Endpoint | Section header; Efficacy<br>Endpoint | There is no primary efficacy endpoint defined in protocol. |
| Section 6.2 | The proportion of subjects in whom the following three conditions are fulfilled at Week 52 (Visit 9): | The proportion of subjects in whom the following three conditions are fulfilled at Week 52 (Visit 9) and at the End of Treatment: | In compliance to<br>Protocol Amendment 3,<br>Version 4.0 |
| Section 6.3 | Section header: Secondary<br>Efficacy Endpoints | Section header: Other<br>Efficacy Endpoints | There is no secondary efficacy endpoints defined in protocol. |
| Section 7.5 | An interim database with a cut off date of December 31, 2011 will be used to provide the NDA safety updates. | An interim study report will<br>be completed to look at<br>safety and efficacy<br>compiled through 31 May<br>2013. | Project team decision. |